CLINICAL TRIAL: NCT06353126
Title: A Prospective, Single Arm, Exploratory Study of Using Drug-eluting Beads Transarterial Chemoembolization Prior to Liver Transplantation in the Treatment of Hepatocellular Carcinoma
Brief Title: DEB-TACE Prior to Liver Transplantation in the Treatment of HCC
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Boston Scientific Corporation (Industry)
Responsible Party: Principal Investigator, Kang He, Professor, RenJi Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DTACELT
Record Dates: First submitted 2024-03-28; First posted 2024-04-08 (Actual); Last update posted 2024-10-18 (Actual); Status verified 2024-10

CONDITIONS: Liver Cancer
MeSH Terms: conditions — Liver Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- DEB-TACE prior to living donor liver transplantation (Experimental): Patients with HCC scheduled for living donor liver transplantation treatment receive DEB-TACE 2 weeks prior to the surgery
  Interventions: Procedure: DEB-TACE

INTERVENTIONS:
Procedure: DEB-TACE — DEB-TACE, or Drug-Eluting Bead Transarterial Chemoembolization, is a minimally invasive interventional radiology procedure primarily used in the treatment of hepatocellular carcinoma (HCC), which is the most common type of liver cancer. This procedure combines two treatment modalities: transarterial chemoembolization (TACE) and the use of drug-eluting beads (DEB).
  During DEB-TACE, tiny beads loaded with chemotherapy drugs are injected directly into the blood vessels supplying the tumor in the liver. These drug-eluting beads gradually release chemotherapy agents, delivering a targeted and sustained dose directly to the cancerous tissue while minimizing systemic side effects. Additionally, the beads themselves act as embolic agents, blocking the blood flow to the tumor and causing ischemia, which further contributes to the destruction of the tumor cells.

SUMMARY:
The goal of the study is to explore whether the usage of DEB-TACE (Drug-Eluting Bead Transarterial Chemoembolization) prior to living donor liver transplantation can prolong the recurrence-free survival in patients with hepatocellular carcinoma (HCC). It is a single-center, exploratory study. The patients scheduled for living donor liver transplantation receive DEB-TACE 2 weeks prior to the surgery.

The primary outcome: Recurrence-free survival (RFS) The secondary outcome:1) Overall survival (OS)；2) Pathological response rate (Pathological Response); 3) Proportion of patients completing living donor liver transplantation; 4) Adverse events related to DEB-TACE.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years;
2. Subjects with viral hepatitis or cirrhosis are clinically diagnosed according to AASLD standards, which require a history of viral hepatitis or cirrhosis combined with imaging examinations (enhanced CT, MRI, second-generation ultrasound contrast agents). When the tumor diameter is greater than 2 cm, a diagnosis can be made if one imaging technique shows typical arterial phase rapid enhancement and rapid washout. If the diameter is 1-2 cm, two imaging techniques must confirm this, or one imaging technique confirms it and alpha-fetoprotein (AFP) is greater than 400 ng/ml. For subjects who cannot be clinically diagnosed, histological or cytological biopsy confirmation is required; original biopsy records can also be used for diagnosis.
3. Child-Pugh score A-B grade;
4. Tumor present in the right lobe of the liver;
5. Liver cancer assessment meeting the "up to seven" criteria: the sum of tumor size and number does not exceed 7;
6. ECOG-PS score 0-1;
7. Scheduled for living donor liver transplantation as the primary treatment;
8. Signed informed consent form.

Exclusion Criteria:

1. Presence of definite cancer thrombi in the main portal vein, vena cava, or main bile duct;
2. Severe hepatic encephalopathy;
3. Coexisting pulmonary arterial hypertension (moderate to high risk, WHO Grade III-IV);
4. Severe contrast agent allergy;
5. Irreversible hepatic artery to hepatic vein shunt;
6. Special types of anatomical variations (Asan portal vein type III);
7. Extrahepatic metastatic tumors;
8. Concurrent active hepatitis or severe infection;
9. Tumor dissemination or distant metastasis, expected survival <3 months;
10. Renal dysfunction, creatinine >176.8 umol/L or creatinine clearance rate <30ml/min;
11. White blood cell count <3.0x109/L, platelet count <50x106/L, and unable to correct;
12. Inability to tolerate surgical anesthesia (severe infection, cardiopulmonary insufficiency, cerebrovascular disease);
13. Severe psychiatric illness;
14. Other reasons deemed unsuitable for participation by the investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2025-07-01 (Estimated); Study Completion 2027-07-01 (Estimated)

PRIMARY OUTCOMES:
Recurrence-free survival (RFS) | 2 years
  the time from DEB-TACE treatment until tumor recurrence in the original site, transplanted liver, other tissues and organs, or death, whichever occurs first.

SECONDARY OUTCOMES:
Overall survival (OS) | 5 years
  the time from DEB-TACE treatment until death from any cause.
Pathological response rate (Pathological Response) | 1 year
  at the time of the surgery
Proportion of patients completing living donor liver transplantation | at the time of the surgery
  1 year
Adverse events related to DEB-TACE | from DEB-TACE to the surgery
  2 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Jianjun Zhang, MD, Principal Investigator — RenJi Hospital
Locations (1):
- Renji Hospital, Shanghai Jiao Tong University School of Medicine, Shanghai, China

IPD SHARING:
Plan to Share IPD: No